CLINICAL TRIAL: NCT01140425
Title: A Phase 1, Randomized, Multiple Dose, Placebo And Active Controlled, 4-Way Crossover Study To Evaluate The Effect Of A Multiple Oral Dose of PF-00232798 On Qt Intervals In Healthy Subjects
Brief Title: Study To Evaluate The Effect Of A Multiple Oral Dose Of PF-00232798 On QT Intervals In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7691017
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: PF-00232798; CCR5; QT; QTc; pharmacokinetics
MeSH Terms: interventions — PF 232798; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-00232798 supratherapeutic dose (Experimental): PF-00232798 supratherapeutic dose
  Interventions: Drug: PF-00232798
- PF-00232798 therapeutic dose (Experimental): PF-00232798 therapeutic dose
  Interventions: Drug: PF-00232798
- Placebo for PF-00232798 (Placebo Comparator): Placebo for PF-00232798
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: PF-00232798 — 600 mg oral solution once daily x 7 days
  Arms: PF-00232798 supratherapeutic dose
Drug: PF-00232798 — 300 mg oral solution once daily x 7 days
  Arms: PF-00232798 therapeutic dose
Drug: Placebo — Oral solution once daily x 7 days
  Arms: Placebo for PF-00232798
Drug: Moxifloxacin — 400 mg tablet single dose
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to assess the affect that PF-00232798 has on QT interval. A prolonged QT interval is a risk factor for arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* 12-lead ECG demonstrating QTc >450 msec at screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* History of orthostatic symptoms or orthostatic hypotension at screening.
* Pregnant or nursing females; females of childbearing potential.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
QTc, using Fridericia's correction method (QTcF) at each time point of PF-00232798 and placebo on Day 7. | 7 days

SECONDARY OUTCOMES:
QTcF, or any other appropriate correction method at each postdose time point of moxifloxacin on Day 7 | 7 days
QTcB or any other appropriate correction method at each postdose time point of PF-00232798 and placebo on Day 7 | 7 days
Pharmacokinetic endpoints for PF-00232798 (Tmax, Cmax, Cτ, and AUClast) | 7 days
Safety and toleration assessed by spontaneous reporting of adverse events, vital signs, 12-lead ECG and laboratory safety assessments | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7691017&StudyName=Study%20To%20Evaluate%20The%20Effect%20Of%20A%20Multiple%20Oral%20Dose%20Of%20PF-00232798%20On%20QT%20Intervals%20In%20Healthy%20Subjects%20